CLINICAL TRIAL: NCT04682015
Title: Effect of a WeChat Platform-based Management Intervention on Blood Pressure Control: A Randomized Clinical Trial.
Brief Title: Effect of a WeChat Platform-based Management Intervention on Blood Pressure Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WMU1H-HTN
Record Dates: First submitted 2020-12-20; First posted 2020-12-23 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2020-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group will be enrolled into WeChat platform. Participants will receive health education materials, monitor blood pressure at home and sent the blood pressure record to the platform and consult doctors online via platform.
  Interventions: Other: WeChat platform group
- Control (No Intervention): Control group will receive usual care and follow up in hospitals and community health centers.

INTERVENTIONS:
Other: WeChat platform group — Participants in the intervention group will receive educational messages related to hypertension, such as impact of hypertension on cardiovascular system, lifestyle adjustment and side effects of antihypertensive drugs. Participants will be reminded to take their blood pressure regularly and enter the blood pressure readings into the WeChat platform. If participants enter extremely high or low readings, they will be asked to seek medical help from doctors. Participants can also consult doctors online via WeChat platform by text and voice messages, or voice calls.
  Arms: Intervention

SUMMARY:
WeChat is the largest and most popular social media platform in China, In this study, investigators will evaluate the use of management program delivered via WeChat platform in patients with hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years with confirmed diagnosis of hypertension
* Office systolic blood pressure (SBP)≥140 mmHg and/or diastolic blood pressure (DBP)≥90 mmHg, or ambulatory blood pressure monitoring (ABPM) indicating 24- hour SBP ≥130 mmHg and/or DBP ≥80 mmHg and/or daytime SBP ≥135 mmHg and/or DBP ≥85 mmHg and/or nocturnal SBP ≥120 mmHg and/or DBP ≥70 mmHg.
* Patients have smart phone and often use WeChat to communicate with others (including written interaction)
* Patients are willing and able to give informed consent for participation in the trial

Exclusion Criteria:

* Secondary hypertension
* Hypertensive emergency: defined as severe elevations in BP (SBP ≥180 mmHg and/or DBP≥120mmHg) associated with evidence of new or worsening target organ damage, including hypertensive encephalopathy, intracranial hemorrhage, cerebral hemorrhage, subarachnoid hemorrhage, cerebral infarction, heart failure, acute coronary syndrome (unstable angina, acute myocardial infarction), aortic dissection, perioperative hypertension, preeclampsia, and eclampsia
* Refractory hypertension: defined as failure to control BP despite lifestyle changes and use of at least 5 antihypertensive agents of different classes, including a thiazide-type diuretic and a mineralocorticoid receptor antagonist
* Pregnancy or lactation or having pregnancy plan during the study period
* Life expectancy less than 1 year
* Participation in another clinical study or clinical trial in the 3 months prior to the confirmation of eligibility or current user of WeChat platform provided by hypertension center of the first affiliated hospital of Wenzhou medical university

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Estimated)
Dates: Start 2021-02-18 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion with controlled blood pressure at 12 months (defined by ambulatory blood pressure monitoring ) | 12 months
  mean 24-hour ambulatory blood pressure monitoring (ABPM) <130/80 mmHg, day time blood pressure <135/85 mmHg, and nocturnal blood pressure <120/70 mmHg

SECONDARY OUTCOMES:
Systolic blood pressure (mmHg) at 12 months | 12 months
  Systolic blood pressure (mmHg) at 12 months
Diastolic blood pressure (mmHg) at 12 months | 12 months
  Diastolic blood pressure (mmHg) at 12 months
Medication adherence at 12 months | 12 months
  Medication adherence will be measured by 8-item self-reported medication-taking scale

CONTACTS AND LOCATIONS:
Overall Officials: GaoJun Wu, Principal Investigator — hypertension center of the first affiliated hospital of Wenzhou medical university